CLINICAL TRIAL: NCT06411379
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Subcutaneous Sonelokimab in Adult Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Study to Evaluate the Efficacy and Safety of Subcutaneous Sonelokimab Compared With Placebo in Adult Participants With Moderate to Severe Hidradenitis Suppurativa
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MoonLake Immunotherapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M1095-HS-302; VELA-2 (Other: Sponsor)
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Hidradenitis; Sweat Gland Diseases; Skin Diseases; Skin Diseases, Bacterial; Suppuration; Anti-Inflammatory Agents; Sonelokimab; Nanobody; Apocrine Gland Disease
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis; Sweat Gland Diseases; Skin Diseases; Skin Diseases, Bacterial; Suppuration | interventions — sonelokimab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- sonelokimab (Experimental): Subjects randomized to this arm will receive sonelokimab 120 mg Q2W from Weeks 0 to 6 then 120 mg Q4W starting at Week 8 up to Week 48.
  Interventions: Drug: Sonelokimab
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo Q2W from Weeks 0 to 6 then Q4W starting at Week 8 up to Week 16. They will receive sonelokimab 120 mg Q2W for 4 doses from Weeks 16 to 22 then Q4W from Week 24 up to Week 48
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sonelokimab — Sonelokimab
  Arms: sonelokimab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a study to evaluate the clinical efficacy and safety of sonelokimab administered subcutaneously compared with placebo in the treatment of adult participants with moderate to severe hidradenitis suppurativa. Participants will be randomized 2:1 to either sonelokimab or matching placebo up to Week 16.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 18 years of age at the time of signing the informed consent.
2. Participants who are diagnosed with hidradenitis suppurativa as determined by the investigator and have a history of signs and symptoms of hidradenitis suppurativa for at least 6 months before signing the informed consent.
3. Participants who have had an inadequate response to appropriate systemic antibiotics for treatment of hidradenitis suppurativa (or demonstrated intolerance to, or had a contraindication to, systemic antibiotics for treatment of their HS), in the investigator's opinion.
4. Participants who have a total AN count of ≥5.
5. Participants who have HS lesions present in ≥2 distinct anatomical areas, at least one of which must contain single or multiple fistulas (ie, be Hurley Stage II or III).

Exclusion Criteria:

1. Participants with a known hypersensitivity to sonelokimab or any of its excipients.
2. Participants with any other active skin disease or condition that may, in the opinion of the investigator, interfere with the assessment of HS.
3. Participants with underlying conditions that, in the opinion of the investigator, potentially places the participant at unacceptable risk.
4. Participants with current severe or uncontrolled disease(s) that put(s) the participant at increased risk in the investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol.
5. Participants with any other known autoimmune disease or any medical condition that in the opinion of the investigator would interfere with an accurate assessment of clinical symptoms of HS.
6. Participants with a gastrointestinal condition including inflammatory bowel disease or diagnosis of ulcerative colitis or Crohn's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-06-17 (Estimated); Study Completion 2026-06-17 (Estimated)

PRIMARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response 75 | Week 16
  Percentage of participants achieving Hidradenitis Suppurativa Clinical Response 75 (HiSCR75), where HiSCR75 is defined as at least a 75% reduction from baseline in abscess and inflammatory nodule (AN) count, with no increase from baseline in abscess or draining fistula count.

SECONDARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response 50 (HiSCR50) | Week 16
  Percentage of participants achieving HiSCR50
Change in International Hidradenitis Suppurativa Severity Score System | Week 16
  Absolute change from baseline in International Hidradenitis Suppurativa Severity Score System (IHS4)
  The IHS4 score is calculated as follows: number of nodules (multiplied by 1) + number of abscesses (multiplied by 2) + number of draining tunnels (multiplied by 4). A total score of 3 or less signifies mild, 4 to 10 signifies moderate, and 11 or higher signifies severe disease.
Dermatology Life Quality Index (DLQI) | Week 16
  Percentage of participants achieving a DLQI total reduction of ≥4 minimal clinically important difference among participants with a baseline DLQI ≥4. DLQI produces a numeric score that can range from 0 to 30. A higher score indicates greater health related quality of life impairment.
Reduction from Numerical Rating Scale (NRS30 & NRS50) in Patient's Global Assessment of Skin Pain (PGA Skin Pain) | week 16
  Percentage of participants achieving at least ≥30% (and ≥50%) reduction and at least 2-unit reduction from Baseline in Numerical Rating Scale (NRS30 & NRS50) in Patient's Global Assessment of Skin Pain (PGA Skin Pain) among subjects with Baseline NRS ≥3
Patient Global Impression - Severity of Illness - Hidradenitis Suppurativa at Week 16 | Week 16
  Percentage of participants with minimal or absent symptoms using the Patient Global Impression - Severity of Illness - Hidradenitis Suppurativa at Week 16. Participants choose the response that best describes the severity of their disease. The question is rated on a 7-point scale ranging from 0 to 6 (0=absent; 1=minimal; 2=mild; 3=moderate; 4=moderately severe; 5=severe; 6=very severe).
Resolution of draining tunnels (DT100) | Week 16 and Week 52
  Percentage of participants with zero draining tunnels in the subgroup of participants with at least one draining tunnel at baseline (DT100)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Kristian Reich, M.D., Ph.D. (equ.), Study Director — MoonLake Immunotherapeutics AG
Locations (95):
- United States (30):
  - Clinical Site, Birmingham, Alabama
  - Clinical Site, North Little Rock, Arkansas
  - Clinical Site, Fountain Valley, California
  - Clinical Site, Santa Monica, California
  - Clinical Site, Aventura, Florida
  - Clinical Site, Hialeah, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Ocala, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, Skokie, Illinois
  - Clinical Site, Plainfield, Indiana
  - Clinical Site, Murray, Kentucky
  - Clinical Site, Baton Rouge, Louisiana
  - Clinical Site, Baltimore, Maryland
  - Clinical Site, Ann Arbor, Michigan
  - Clinical Site, Canton, Michigan
  - Clinical Site, Clarkston, Michigan
  - Clinical Site, Waterford, Michigan
  - Clinical Site, New Brighton, Minnesota
  - Clinical Site, Omaha, Nebraska
  - Clinical Site, Las Vegas, Nevada
  - Clinical Site, New York, New York
  - Clinical Site, Fargo, North Dakota
  - Clinical Site, Columbus, Ohio
  - Clinical Site, Murfreesboro, Tennessee
  - Clinical Site, Dallas, Texas
  - Clinical Site, Plano, Texas
  - Clinical Site, San Antonio, Texas
  - Clinical Site, Morgantown, West Virginia
  - Clinical Site, Milwaukee, Wisconsin
- Belgium (4):
  - Clinical Site, Ghent
  - Clinical Site, Leuven
  - Clinical Site, Liège
  - Clinical Site, Woluwe-Saint-Lambert
- Bulgaria (2):
  - Clinical Site, Sofia
  - Clinical Site, Stara Zagora
- Canada (8):
  - Clinical Site, Calgary, Alberta
  - Clinical Site, Edmonton, Alberta
  - Clinical Site, Guelph, Ontario
  - Clinical Site, Peterborough, Ontario
  - Clinical Site, Richmond Hill, Ontario
  - Clinical Site, Toronto, Ontario
  - Clinical Site, Windsor, Ontario
  - Clinical Site, Saskatoon, Saskatchewan
- Czechia (2):
  - Clinical Site, Ostrava
  - Clinical Site, Prague
- France (11):
  - Clinical Site, Antony
  - Clinical Site, Besançon
  - Clinical SIte, Brest
  - Clinical Site, Dijon
  - Clinical Site, Le Mans
  - Clinical Site, Lyon
  - Clinical Site, Montpellier
  - Clinical Site, Rouen
  - Clinical Site, Saint-Mandé
  - Clinical Site, Saint-Priest-en-Jarez
  - Clinical Site, Toulouse
- Germany (13):
  - Clinical Site, Augsburg
  - Clinical Site, Bad Bentheim
  - Clinical Site, Berlin
  - Clinical Site, Bielefeld
  - Clinical Site, Bochum
  - Clinical Site, Bramsche
  - Clinical Site, Darmstadt
  - Clinical Site, Dresden
  - Clinical Site, Gera
  - Clinical Site, Hamburg
  - Clinical Site, Kiel
  - Clinical Site, Lübeck
  - Clinical Site, Würzburg
- Clinical Site, Dublin, Ireland
- Clinical Site, Rotterdam, Netherlands
- Poland (8):
  - Clinical Site, Chorzów
  - Clinical Site, Katowice
  - Clinical Site, Kielce
  - Clinical Site, Olsztyn
  - Clinical Site, Poznan
  - Clinical Site, Szczecin
  - Clinical Site, Warsaw
  - Clinical Site, Wroclaw
- Clinical Site, Trnava, Slovakia
- Spain (14):
  - Clinical Site, Alcorcón
  - Clinical Site, Alicante
  - Clinical Site, Badalona
  - Clinical Site, Barcelona
  - Clinical Site, Cadiz
  - Clinical Site, Córdoba
  - Clinical Site, Granada
  - Clinical Site, Granollers
  - Clinical Site, Madrid
  - Clinical Site, Manises
  - Clinical Site, Málaga
  - Clinical Site, Santiago de Compostela
  - Clinical Site, Seville
  - Clinical Site, Valencia